CLINICAL TRIAL: NCT05676710
Title: A Single-arm, Open-label, Pilot Study on the Efficacy and Safety of PI3K Inhibitors in Relapsed/Refractory Large Granular T Lymphocytic Leukemia
Brief Title: Efficacy and Safety of PI3K Inhibitors in Relapsed/Refractory Large Granular T Lymphocytic Leukemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Collaborators: YL-Pharma (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT2022068
Record Dates: First submitted 2022-12-08; First posted 2023-01-09 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2023-12

CONDITIONS: Relapsed/Refractory Large Granular T Lymphocytic Leukemia
MeSH Terms: conditions — Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): PI3K inhibitors
  Interventions: Drug: Linperlisib

INTERVENTIONS:
Drug: Linperlisib — Elevated PI3K activity in T-LGL likely plays an important role in the ability of the pathologic cells to avoid homeostatic apoptosis, since inhibition of this pathway leads to apoptosis in the population of cells harboring the pathologic clone. More importantly, the activity of this pathway may represent a kind of "Achilles heel" for T-LGL in that PI3K inhibitors alone are quite effective at inducing spontaneous apoptosis in the clonal CTLs after a short incubation.

SUMMARY:
This is a prospective, multicenter, single-arm, pilot study. The aim of this study is to evaluate the efficacy and safety of linperlisib, the PI3K delta inhibitor for patients with relapsed/refractory large granular T lymphocytic leukemia.

ELIGIBILITY:
Inclusion Criteria:

* Male or female age ≥ 18 years
* Diagnosis of T-cell large granular lymphocytic leukemia (T-LGLL)
* Meet any of the following indications for treatment：

  1. Hemoglobin < 100g/L or RBC transfusion dependence
  2. Neutrophil count <0.5×10^9/L or neutrophil count decreased with recurrent infection
  3. Progressive splenomegaly and/or Massive Splenomegaly
  4. Combined with autoimmune diseases requiring treatment, such as rheumatoid arthritis, autoimmune thyroiditis, etc.
  5. Severe B symptoms
* Failure or intolerance to a first-line therapy
* ECOG performance status ≤2
* Expected survival ≥ 6 months
* Willing and able to comply with the requirements for this study and written informed consent.

Exclusion Criteria:

* History of other lymphoproliferative neoplasms
* Had malignant tumor within 5 years before enrollment, exclusive of cured basal or squamous cell skin cancer, superficial bladder cancer, prostate intraepithelial tumor, cervical carcinoma in situ or other indolent tumors
* Previously received organ or stem cell transplantation.
* Patients with active infection within 2 weeks before giving the first dose of medication
* Patients with HBV, HCV, HIV or other infections that require treatment
* History of immunodeficiency, or congenital immunodeficiency disorders
* Any severe and/or uncontrolled medical conditions or other conditions that could affect their participation in the study, including clinically significant cardiac diseases, refractory hypertension, metabolic disorders and other diseases that seriously affect the function of the gastrointestinal tract.
* Abnormal liver function: two consecutive examinations with an interval of ≥1 week suggest that ALT and AST are 2.5 times higher than the upper limit of normal values
* Renal impairment: creatinine clearance <60ml/min
* History of pulmonary fibrosis, interstitial pneumonia, pneumoconiosis, radiation pneumonitis, drug-related pneumonia, severe impairment of lung function, etc.
* Received attenuated vaccine 4 in weeks before enrollment
* Participation in another clinical trial within 4 weeks before the start of this trial
* Have an allergy to Linperlisib or any other part of this medicine.
* Previously treated with other PI3Kδ inhibitor.
* Pregnant or breast-feeding patients
* Patients considered to be ineligible for the study by the investigator for reasons other than the above

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2023-02-10 (Actual); Primary Completion 2024-01-30 (Actual); Study Completion 2024-02-14 (Actual)

PRIMARY OUTCOMES:
Overall response rate: HPR + HCR + CMR | 8 weeks
  Percentage of patients with hematological response. Hematological response is evaluated by hemoglobin (Hb), absolute neutrophil count (ANC), platelet count (PLT), absolute lymphocyte count (ALC), absolute large granular lymphocyte count, and blood transfusion.

SECONDARY OUTCOMES:
Incidence of the adverse event | 8 weeks
  Use Common Terminology Criteria for Adverse Events (CTCAE) Version 5 to assess the adverse event
Time to achieve partial hematologic response (HPR) | 8 weeks
  Duration time was calculated from enrollment to achieve HPR. HPR is assessed by Hb, ANC, PLT, ALC, absolute large granular lymphocyte count and blood transfusion
Time to achieve complete hematologic response (HCR) | 8 weeks
  Duration time was calculated from enrollment to achieve HCR. HCR is assessed by Hb, ANC, PLT, ALC, and absolute large granular lymphocyte count.
Time to achieve complete molecular response (CMR) | 8 weeks
  Duration time was calculated from enrollment to achieve CMR. CMR is assessed by Hb, ANC, PLT, ALC, and absolute large granular lymphocyte count
Change of the health-related quality of life | Baseline and 2 cycles of therapy
  Medical Outcomes Study Questionnaire Short Form 36 Health Survey (SF-36) is used to assess the health-related quality of life of patients. The SF-36 has eight scaled scores; the scores are weighted sums of the questions in each section. Scores range from 0 - 100. Lower scores = more disability, higher scores = less disability
Relapse free survival (RFS) | A minimum of 2 years of planned follow-up
  Duration time was calculated from response to relapse.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Zhoukou Central Hospital, Zhoukou, Henan
  - Regenerative Medicine Center, Tianjin, Tianjin Municipality

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhang L, Qiu C, Li R, Shen Y, Tian L, Chang H, Liang Q, Pan H, Gao Z, Li W, Zhao J, Fang L, Yu X, Xu J, Kuang Z, Yuan W, Chu Y, Shi J. KLRG1 re-defines a leukemic clone of CD8 effector T cells sensitive to PI3K inhibitor in T cell large granular lymphocytic leukemia. Cell Rep Med. 2025 Apr 15;6(4):102036. doi: 10.1016/j.xcrm.2025.102036. Epub 2025 Mar 26. PMID 40147444